CLINICAL TRIAL: NCT00743314
Title: Integration of SPECT/CT Lymphoscintigraphy Into Breast Cancer Radiation for LymphaticSparing
Brief Title: Single-Photon Emission Computed Tomography, Computed Tomography Lymphoscintigraphy, and Intensity-Modulated Radiation Therapy in Treating Patients Who Have Undergone Surgery for Stage I or Stage II Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000611987; P30CA015083 (NIH); MC0734 (Other: Mayo Clinic Cancer Center); 07-008292 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Lymphedema
Keywords: lymphedema; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Radiotherapy, Intensity-Modulated; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: screening questionnaire administration
Procedure: computed tomography
Procedure: lymphoscintigraphy
Procedure: single photon emission computed tomography
Radiation: intensity-modulated radiation therapy
Radiation: technetium Tc 99m sulfur colloid

SUMMARY:
RATIONALE: Diagnostic procedures, such as single-photon emission computed tomography and computed tomography lymphoscintigraphy, may help lower the dose of radiation therapy after surgery, and help prevent lymphedema.

PURPOSE: This clinical trial is studying single-photon emission computed tomography and computed tomography lymphoscintigraphy followed by intensity-modulated radiation therapy to see how well they work in treating patients who have undergone surgery for stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the feasibility of integrating Philips Precedence SPECT/CT® images with GE PET/CT Fusion software to reduce radiation dosimetry delivered to lymph nodes draining the arm in patients after surgery for stage I or II breast cancer.
* To examine the differences in radiation dosimetry in these patients using 3-D conformal radiotherapy with vs without the Philips Precedence SPECT/CT®.
* To compare reduction in lymph node radiation dosimetry in these patients using single photon emission computed tomography (SPECT) and computed tomography (CT) with 3-D conformal radiotherapy vs intensity-modulated radiotherapy.

OUTLINE: Patients receive filtered technetium Tc 99m sulfur colloid (TcSC) intradermally and undergo single photon emission computed tomography (SPECT) and computed tomography (CT) imaging at the time of TcSC and 2 hours after injection. Patients then undergo intensity-modulated radiotherapy of the whole breast, including the low axilla and lymph nodes identified by the Phillips Precedence SPECT/CT® at a dose determined by computer analysis of the imaging information.

Patients complete a lymphedema screening questionnaire at baseline and at 12 and 24 months after treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven primary invasive breast cancer, meeting one of the following criteria:

  * Stage I or II disease with negative sentinel or axillary node dissections
  * Stage II disease with micrometastases (defined as < 2.0 mm focus) in 1-2 lymph nodes and/or a single positive axillary node ≤ 1 cm with no extracapsular extension
* Completed all surgical intervention (e.g., lumpectomy, mastectomy)
* Planning adjuvant whole breast irradiation including the low axilla
* No bilateral or recurrent breast cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnancy or nursing
* Negative pregnancy test
* Able to complete questionnaire(s) alone or with assistance
* No active infection
* No history of invasive cancer within the past 5 years, except basal cell or squamous cell skin cancers

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior surgery or radiation to the ipsilateral breast or axilla
* No concurrent neoadjuvant chemotherapy or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Philips Precedence SPECT/CT® and GE PET/CT Fusion software integration
Dosimetry differences between 3-D conformal radiotherapy with vs without the Philips Precedence SPECT/CT®
Lymph node dosimetry differences between single photon emission computed tomography (SPECT) and computed tomography (CT) with 3-D conformal radiotherapy vs intensity-modulated radiotherapy
Association between radiation exposure and limb volume, circumferential wrist measurements, circumferential forearm measurements, and extra-cellular fluid measurements

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Cheville, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States